CLINICAL TRIAL: NCT05952479
Title: Handgrip Strength, Lean Mass, and Blood Pressure in Primary School Children Aged 8-10 Years Old With Undernutrition
Brief Title: The Comparison of Handgrip Strength, Lean Mass, and Blood Pressure in Primary School Children Aged 8-10 Years Old With Undernutrition and Normal Nutritional Status
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitas Airlangga (Other)
Collaborators: Indonesia University (Other); Gadjah Mada University (Other); Lembaga Pengelola Dana Pendidikan (Indonesia Endowment Fund for Education) (Unknown)
Responsible Party: Principal Investigator, Nur Aisiyah Widjaja, Principal Investigator and Medical Staf in Pediatric Nutrition and Metabolic Disease, Universitas Airlangga
Other Study IDs: Third ID
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Undernutrition
Keywords: Handgrip strenght; Undernutrition; Nutritional status
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Undernutrition: Undernutrition is defined as weight-for-age z-score (WAZ), height-for-age z-score (HAZ), and weight-for-height z-score (WHZ) of WHO growth chart standards < -2.00 SD
- Normal nutrition: Normal nutrition is defined as weight-for-age z-score (WAZ), height-for-age z-score (HAZ), and weight-for-height z-score (WHZ) of WHO growth chart standards in the range of +2 and -2.00 SD

SUMMARY:
Undernutrition occurs in 900 million individuals globally, so it is a very important health problem because it contributes to high mortality rates, especially in children. In addition, undernutrition has consequences for children's growth and development, including increased susceptibility to 1) Experiencing fat accumulation, especially in the central part of the body; 2) Experiencing changes in body metabolism, especially fat, decreased oxidation; 3) Experiencing a decrease in resting energy expenditure and postprandial energy expenditure; 4) Insulin resistance in adulthood which results in hypertension and dyslipidemia, 5) Decreased capacity to do manual work that requires physical strength. 6) Changes occur in the function of the autonomic nervous system (Matrins et al., 2011). Loss of muscle mass and function causes muscle weakness. Handgrip strength has been used as a tool to measure muscle strength and functionality and can measure low individual mobility because handgrip strength is positively correlated with daily activity (Whiting et al., 2016). Hand grip strength or handgrip strength is used as a predictor of undernutrition in adult patients with cancer who are hospitalized (Bauer et al., 2015), and is stated as a predictor of nutritional status and changes in nutritional status (Flood et al., 2014). Other research also shows that there is a positive correlation between BMI percentile and hand grip strength (Kotecha and Desai, 2022). In studies on elderly populations, handgrip strength is positively correlated with nutritional status (Akbar and Setiati, 2018), while in populations of children at risk of malnutrition (using the Paediatric Yorkhill Malnutrition Score-PYM), it shows handgrip strength based on age (HGS z-score). and based on height is lower than children who have a lower risk of malnutrition. The HGS z-score can also be used as a predictor of fat free mass (FFM) for sick children compared to healthy children and is also related to plasma CRP (Mckirdy et al., 2021).

Based on the explanation above, this research was conducted to know the differences in hand grip strength, muscle mass, and blood pressure in undernourished children aged 8-10 years compared to normal children.

DETAILED DESCRIPTION:
An experimental study with an analytic cross-sectional design examines muscle mass, hand grip strength, and blood pressure in children with undernutrition compared to normal. The subjects are elementary school children aged 8-10 years with undernutrition and overnutrition. Undernutrition was determined after measuring body weight and height, then weight/age, height/age, and weight/height z-scores were determined using the WHO Anthroplus software. If < -2 SD, then grouped into undernutrition, but if 0 to -2 SD then grouped into normal. Homogeneity and normality tests were carried out on the variables age, weight, height, anthropometry, arm and waist circumference, hand grip strength, muscle mass, and blood pressure. Data is presented in descriptive form (x + SD). A paired sample t-test (or Mann-Whitney test) was performed on these variables, dividing the subjects into 2: undernutrition vs. normal, with significance >0.05. Relationships between variables were analyzed using Pearson's or Spearman's correlation.

1. After obtaining permission and approval from the school, the researcher conducted an initial screening by measuring height and weight, as well as the age of the prospective subject/
2. Determination of nutritional status using WHO Anthroplus to determine undernourished and normal nutritional subjects
3. Furthermore, the researchers reported the findings to the school for socialization and the signing of informed consent by parents
4. Researchers re-measurement of weight, height, waist circumference, blood pressure and handgrip strength in subjects who are willing to take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 years until 10 years
* Study in Primary School in Surabaya
* Healthy
* Volunteer to participate in this study (the parents sign the informed consent we sent)

Exclusion Criteria:

* Had autoimmune disease, congenital disorders, or other chronical disease
* Retire during the observational periods
* Consumed steroids, antibiotics or hormone therapy

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects are elementary school children aged 8-10 years with undernutrition and overnutrition. Undernutrition was determined after measuring body weight and height, then weight/age, height/age and weight/height z-scores were determined using the WHO anthroplus software. If < -2 SD, then grouped into undernutrition, but if 0 to -2 SD then grouped into normal.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Body weight | 1 year
  Body weight will be measured using Tanita RD 953-BK digital scale (presenting in mean +/- SD, in kg). The subjects were asked to step at the scale in an upright state. The body weight appears on the screen and is then noted in the data collection sheet. The subject must use light clothes without accessories or footwear
Body height | 1 year
  Body height will be measured using a stadiometer Seca 213 (presenting in mean +/- SD, in cm). The subjects were asked to stand upright on the stadiometer base, with the heel, buttock, and shoulder blades touching the scale pool, their chin up, look straight ahead. The head slider was lowered until it touched the cranium. The body height was noted on the data collection sheet.
Blood pressure | 1 year
  Blood pressure will be measured using Omron Automatic Blood Pressure Monitor (Omron Health Care Co., Ltd, Japan) (in mmHg), by placing the cuff on the right arm, then pulling and tightening it according to the size of the arm. After it was installed correctly (fasten and did not move), the power button on the digital tension tool was pressed, and then the microprocessor started to drive air pressure into the cuff, and then the value of blood pressure will appear in the manometer tube column. Blood pressure measurement was performed in a sitting position after the subject had rested for 10 minutes. The data will be presented as mean +/- standard deviation (SD)
Handgrip strength | 1 year
  Handgrip strength will be measured using handgrip dynamometry (Camry) Patients sat comfortably on a chair and, after adjusting the handle of the dynamometer, patients were advised to hold the instrument away from the body and table. Patients were then advised to hold and compress the handle of the dynamometer with as much strength as possible with the dominant hand. Three readings were noted with a gap of more than 30 seconds. The mean of the 3 recordings was taken into consideration. Data presented as mean +/- SD, in kg

CONTACTS AND LOCATIONS:
Locations (1):
- SDN Airlangga III, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The data will be shared in Airlangga Repository